CLINICAL TRIAL: NCT05354076
Title: Study on the Correlation Between Immunoglobulin and Liposomal Doxorubicin in Vivo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-liposomal doxorubicin-01
Record Dates: First submitted 2021-12-22; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liposomal doxorubicin (Experimental): According to the clinical diagnosis and treatment norms, it is suitable for patients with advanced malignant tumors diagnosed by histopathology with doxorubicin hydrochloride liposome injection chemotherapy.
  Interventions: Drug: doxorubicin hydrochloride liposome injection

INTERVENTIONS:
Drug: doxorubicin hydrochloride liposome injection — According to the clinical diagnosis and treatment norms, it is suitable for patients with advanced malignant tumors diagnosed by histopathology with doxorubicin hydrochloride liposome injection chemotherapy.(For breast cancer patients: liposomal doxorubicin 35mg/m2 q3w)

SUMMARY:
To study the correlation between the content of natural IgM in patients' blood samples and liposomal doxorubicin for clinical use, and to explore the possibility of using natural IgM content to guide clinical accurate medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years (including cutoff value), regardless of gender.
2. According to the clinical diagnosis and treatment norms, it is suitable for patients with advanced malignant tumors diagnosed by histopathology with doxorubicin hydrochloride liposome injection chemotherapy.
3. Eastern Cooperative Oncology Group Performance Status of 0-1.
4. Life expectancy ≥ 3 months.
5. Adequate function of major organs meets the following requirements :

   1. Neutrophils ≥ 1.5×10^9/L
   2. Platelets ≥ 75×10^9/L
   3. Hemoglobin ≥ 90g/L
   4. Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
   5. ALT and AST ≤ 2.5 × ULN, Subjects with liver metastasis require TBIL ≤ 1.5 × ULN, ALT and AST ≤ 5 × ULN。
   6. BUN and Cr ≤ 1.5 × ULN, Or creatinine clearance (CCR) ≥ 50 ml / min.
   7. International normalized ratio(INR)≤1.5 × ULN，activated partial thromboplastin time(APTT) ≤ 1.5 × ULN
6. Women should agree to use effective contraceptives (such as intrauterine device [IUD], contraceptive or condom) during the study period and within 6 months after the end of the study; serum pregnancy test is negative within 7 days before the study and must be non lactating subjects; men should be the same subjects who intend to use contraceptives during the study period and within 6 months after the end of the study period.
7. Patients volunteered to participate in the study, signed informed consent, and were able to follow the blood sampling, visit and related procedures specified in the trial.

Exclusion Criteria:

1. Received systemic therapy such as chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatments within 4 weeks before enrollment; according to the judgment of the researcher, the cleaning period can be appropriately shortened or extended. For example, for endocrine drugs, in order to avoid making patients wait too long, the cleaning period can be appropriately shortened to 2 weeks.
2. Those weighing less than 40 kg.
3. Previously received any liposomal doxorubicin analogues treatment.
4. Patients with a history of allergy to liposomes or adriamycin.
5. Have a history of serious cardiovascular disease, such as severe cardiac rhythm or conduction abnormalities (ventricular arrhythmia requiring clinical intervention, degree II ~ III atrioventricular block, etc.), cardiac infarction, history of coronary artery bridging surgery, heart failure, NYHA grade II or above, left ventricular ejection fraction (LVEF) ≤ 50%, male QTCF > 450msec or female QTCF > 470msec, etc.
6. Patients with active infection (NCI CTC AE v5.0 ≥ grade 2).
7. Patients have a history of autoimmune diseases and immune defects, including HIV test positive, or have other acquired and congenital immune defects, or have a history of organ transplantation and need to take corticosteroids routinely.
8. Hepatitis B surface antigen positive (HBsAg), and peripheral blood hepatitis B virus DNA (HBV-DNA) titer detection is more than 1. ×103 IU / ml; If HBsAg is positive and HBV-DNA in peripheral blood is less than 1 × 103IU/mL, if the researchers believe that the chronic hepatitis B is stable and does not increase the risk of the subjects, the subjects are eligible to be selected.
9. Anti hepatitis C virus antibody and anti treponema pallidum specific antibody were positive.
10. Have a clear history of neurological or mental disorders, including epilepsy or dementia.
11. Patients with clinical symptoms of central nervous system metastasis or meningeal metastasis, or other evidence indicating that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, patients with asymptomatic brain metastasis, or stable clinical symptoms without steroid hormone and other treatment for brain metastasis for ≥ 28 days can be enrolled.
12. According to the judgment of the investigator, there are other accompanying diseases that seriously endanger the safety of the patient or affect the completion of the study.
13. Pregnant or lactating female subjects.
14. Patients considered unsuitable by the investigator to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2000-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The content of natural IgM in patients' blood samples | 6 weeks
  IgM regulates the performance of liposomes by regulating the efficiency of liposomes activating complement in vivo. Among many immunoglobulins, IgM rather than IgG is the key plasma protein affecting the efficiency of liposomes activating complement.The content of IgM in serum were detected by ELISA
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0 | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China